CLINICAL TRIAL: NCT01122524
Title: A Prospective, Multi-center Observational Study With Blinded, Nested Case:Control Analyses to Evaluate the Performance of the Verinata Health Prenatal Aneuploidy Diagnostic Test
Brief Title: MatErnal BLood IS Source to Accurately Diagnose Fetal Aneuploidy
Acronym: MELISSA
Status: Completed | Type: Observational
Sponsor: Verinata Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ART-0006
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Pregnant Women; Prenatal Care
Keywords: Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chromosomal Abnormality: Fetus affected by chromosomal abnormality
- No Chromosomal Abnormality: Fetus not affected by chromosomal abnormality

SUMMARY:
The primary objective of this study is to determine the performance characteristics (sensitivity and specificity) of the Verinata Health Test to detect fetal Trisomy 21 (T21) compared to karyotype results obtained by amniocentesis or chorionic villus sampling (CVS).

Secondary objectives are to assess performance of the test to detect male gender (XY) and other less common aneuploidies (Trisomy 13 (T13), Trisomy 18 (T18), and Turner Syndrome (45, X)) compared to clinical fetal karyotype.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinically confirmed viable pregnancy at the time of enrollment
* Clinically determined gestational age between 8 wks, 0 days and 22 wks, 0 days
* Referred or planning to undergo CVS or amniocentesis procedure due to risk of fetal aneuploidy based on protocol-specified clinical indicators
* Able to provide consent for participation using language appropriate forms and consent process

Exclusion Criteria:

- Invasive prenatal procedure (amniocentesis or CVS) performed prior to enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women undergoing chorionic villus sampling (CVS) or amniocentesis
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Classification of fetal status as affected or not affected for Trisomy 21 based on Artemis Health Test on maternal blood. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Sehnert, MD, Study Director — Verinata Health, Inc.
Locations (11):
- United States (11):
  - Center for Fetal Medicine, Los Angeles, California
  - San Francisco Perinatal Associates, San Francisco, California
  - Women's Clinic of Northern Colorado, Fort Collins, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - OB/Gyn Specialists of the Palm Beaches, West Palm Beach, Florida
  - New Mexico Consortium for Perinatal Research, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - The Women's Hospital of Texas, Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Background] http://www.clinchem.org/cgi/content/abstract/clinchem.2011.165910
- [Derived] Bianchi DW, Prosen T, Platt LD, Goldberg JD, Abuhamad AZ, Rava RP, Sehnert AJ; MatErnal BLood IS Source to Accurately diagnose fetal aneuploidy (MELISSA) Study Group*. Massively parallel sequencing of maternal plasma DNA in 113 cases of fetal nuchal cystic hygroma. Obstet Gynecol. 2013 May;121(5):1057-1062. doi: 10.1097/AOG.0b013e31828ba3d8. PMID 23635743
- [Derived] Bianchi DW, Platt LD, Goldberg JD, Abuhamad AZ, Sehnert AJ, Rava RP; MatErnal BLood IS Source to Accurately diagnose fetal aneuploidy (MELISSA) Study Group. Genome-wide fetal aneuploidy detection by maternal plasma DNA sequencing. Obstet Gynecol. 2012 May;119(5):890-901. doi: 10.1097/AOG.0b013e31824fb482. PMID 22362253